CLINICAL TRIAL: NCT02396732
Title: The Role Of Combined Therapy With Aspirin and Enoxaparin In Prevention Of Venous Thromboembolism In Trauma Patients: A Randomized-Controlled Trial
Brief Title: Aspirin and Enoxaparin for VTE in Trauma
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated due to futility and less subjects meeting entry criteria
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Kenneth Proctor, Professor of Surgery, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20140937
Record Dates: First submitted 2015-03-12; First posted 2015-03-24 (Estimated); Results first posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-10

CONDITIONS: Venous Thromboembolism; Thromboprophylaxis; Trauma
Keywords: Aspirin; Enoxaparin; Thromboprophylaxis; Trauma; Venous thromboembolism
MeSH Terms: conditions — Venous Thromboembolism; Wounds and Injuries | interventions — Aspirin; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Molecular Weight Heparin (LMWH) + Aspirin (ASA) (Experimental): Group will get both enoxaparin (standard of care) and aspirin (intervention) after consent up to Intensive Care Unit (ICU) discharge.
  Interventions: Drug: Aspirin; Drug: Enoxaparin
- Low Molecular Weight Heparin (LMWH) Alone (Active Comparator): Group will get only enoxaparin (standard of care) after consent up to Intensive Care Unit (ICU) discharge.
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Aspirin — Daily dose is 81 mg oral tablet
  Arms: Low Molecular Weight Heparin (LMWH) + Aspirin (ASA)
Drug: Enoxaparin — Daily dose is by subcutaneous injection and weight based at the discretion of the treating clinician.

SUMMARY:
The purpose of this study is to determine if the addition of antiplatelet therapy (i.e. aspirin) to low-molecular-weight-heparin (i.e. enoxaparin) will decrease the incidence of venous thromboembolism (VTE) in high-risk critically injured patients. The investigators further aim to determine the safety and efficacy of dual thromboprophylaxis with aspirin and enoxaparin for decreasing the incidence of VTE after trauma.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Blunt or penetrating trauma
* Requires VTE thromboprophylaxis
* High-risk for VTE

Exclusion Criteria:

* Presence of VTE upon admission
* Pregnant or nursing
* Inability to give informed consent by patient or healthcare proxy
* Contraindication to enoxaparin
* Contraindication to aspirin
* Epidural or subdural hematoma
* Presence, or removal within the last 12 hours, of an epidural or spinal catheter, or recent (within the last 12 hours) epidural or spinal anesthesia/procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-02; Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Proctor, PhD, Principal Investigator — University of Miami
Locations (1):
- Ryder Trauma Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- LMWH + ASA: Group will get both enoxaparin (standard of care) and aspirin (intervention) after consent up to Intensive Care Unit (ICU) discharge.
- LMWH Alone: Group will get only enoxaparin (standard of care) after consent up to Intensive Care Unit (ICU) discharge.
Period: Overall Study
Arm/Group | LMWH + ASA | LMWH Alone
Started | 14 | 17
Completed | 14 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LMWH + ASA | LMWH Alone | Total
Number analyzed (Participants) | 14 | 17 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (13) | 40 (16) | 40 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 11 | 11 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3 | 7 | 10
  Hispanic / Latino | 8 | 8 | 16
  White | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Venous Thromboembolism
Description: Incidence of VTE is defined as new cases reported of: 1. Deep Vein Thrombosis (DVT), symptomatic or asymptomatic as assessed via venous duplex ultrasonography, and 2. Pulmonary Embolism (PE), symptomatic or asymptomatic as assessed via chest computed tomography with angiography (CTA) or ventilation-perfusion (VQ) Scan
Time Frame: Up to 2 months of hospitalization
Measure: Number; unit: incidents
Arm/Group | LMWH + ASA | LMWH Alone
Number analyzed (Participants) | 14 | 17
incidents | 1 | 3

2. Secondary Outcome: Change in Hypercoagulability
Description: Assessed via the combination of routine laboratory values (Prothrombin Time and Partial Thromboplastin Time) evaluated through weekly thromboelastography (TEG)
Time Frame: Baseline, up to 2 months hospitalization
Population: Data analysis was not completed for this outcome as samples were not collected as per protocol.
Arm/Group | LMWH + ASA | LMWH Alone
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Mortality
Description: Mortality will be reported as the number of participants with reported death upon hospital discharge
Time Frame: Up to 2 months of hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | LMWH + ASA | LMWH Alone
Number analyzed (Participants) | 14 | 17
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 2 months
Description: For purposes of this study we are only collecting and reporting the following adverse events: Acute Respiratory Syndrome, Altered Mental Status, Bacteremia, Pneumonia, Venous Thromboembolism, Bleeding Complications, Acute Kidney Injury, Urinary Tract Infection, Surgical Site Infection and Mortality.
Arm/Group | LMWH + ASA | LMWH Alone
All-Cause Mortality (participants affected / at risk) | 0/14 | 1/17
Serious Adverse Events (participants affected / at risk) | 2/14 | 4/17
Other Adverse Events (participants affected / at risk) | 1/14 | 1/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LMWH + ASA (N=14) | LMWH Alone (N=17)
Altered Mental Status (General disorders) | 1 (1) | 0 (0)
Venous Thromboembolism (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Bacteremia (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LMWH + ASA (N=14) | LMWH Alone (N=17)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT02396732/Prot_SAP_000.pdf